CLINICAL TRIAL: NCT06060678
Title: Evaluation of the Efficacy of Genicular Nerve Alcohol Neurolysis in the Management of Knee Osteoarthritis Pain
Brief Title: Efficacy of Genicular Nerve Alcohol Neurolysis in Knee Osteoarthritis Pain
Status: Completed | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Medical doctor, Diskapi Teaching and Research Hospital
Other Study IDs: Genicular alcohol neurolysis
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Knee Pain Chronic
Keywords: Osteoarthritis; Pain; Ultrasonography; Paresthesia
MeSH Terms: conditions — Osteoarthritis; Pain; Paresthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to evaluate the efficacy of genicular nerve alcohol neurolysis in the treatment of pain caused by chronic knee osteoarthritis. The investigators will evaluate the efficacy of genicular nerve alcohol neurolysis using the numeric rating scale (NRS) and the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). NRS and WOMAC scores will be evaluated before, 1, and 3 months after the procedure.

DETAILED DESCRIPTION:
Alcohol neurolysis of the genicular nerve is a procedure that involves injecting alcohol around the nerve branches that supply sensation to the knee joint. The alcohol destroys the nerve fibers and blocks the transmission of pain signals from the knee to the brain. This technique can be used to treat chronic knee pain caused by osteoarthritis (OA).

Several studies have reported that alcohol neurolysis of the genicular nerve can provide significant pain relief and functional improvement in patients with knee OA or postoperative pain. For example, Dass et al. (1) reported two cases of alcohol neurolysis of the genicular nerve using fluoroscopy and ultrasonography in patients with knee OA or persistent postsurgical pain of the knee. Both patients had more than 50% reduction in their numerical rating scale (NRS) scores and improved range of motion and quality of life at 3 months follow-up.

Ultrasonography-guided genicular nerve alcohol neurolysis is prominent with its easy applicability and low cost. There are no studies in the literature evaluating the efficacy of genicular nerve alcohol neurolysis for chronic knee OA. In this prospective study, the investigators will evaluate the NRS and WOMAC scores of patients who underwent genicular nerve alcohol neurolysis for chronic knee OA before, 1, and 3 months after the procedure. In addition, the incidence of procedure-related adverse events (such as paresthesia) recorded in patient records will be analyzed.

1. Dass RM et al. Alcohol neurolysis of genicular nerve for chronic knee pain. Korean J Pain 2019; 32 (3): 223-227. https://www.epain.org/journal/view.html?doi=10.3344/kjp.2019.32.3.223

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe knee pain due to knee osteoarthritis (0-10 pain of intensity 6 and above on an inter-numeric pain scale)
* Permanent pain for more than 6 months
* Grade 3 or 4 in the radiological Kellgren-Lawrence classification having osteoarthritis
* Pain with conservative methods such as analgesics and physiotherapy treatment failure

Exclusion Criteria:

* History of intra-articular knee intervention in the last 6 months
* Cognitive impairment
* Hepatic or renal insufficiency
* Severe psychiatric illness
* Local or systemic infection
* Coagulopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients who underwent genicular nerve alcohol neurolysis for knee osteoarthritis pain
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-05 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) | Change from Baseline NRS at 1 and 3 months
  Patients are asked to circle the number between 0 and 10, 0 and 20 or 0 and 100 that fits best to their pain intensity.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Change from Baseline WOMAC at 1 and 3 months
  The WOMAC Pain score ranges from 0 to 20 with higher scores equating to greater pain with activities of daily living. The generic pain scale ranges from 0 to 10 for the OAI and 0 to 100 for MOST, with higher scores equating to greater pain

CONTACTS AND LOCATIONS:
Overall Officials: Gevher Rabia Genc Perdecioğlu, Study Chair — Diskapi TRH
Locations (1):
- Diskapi Training and Research Hospital, Ankara, Turkey (Türkiye)